CLINICAL TRIAL: NCT03292250
Title: Public-interest Multicenter Umbrella Trial Based on Genetic Analysis in Korean Head and Neck Cancer and Esophageal Cancer Patient - Part 1 (HNSCC)]
Brief Title: Korean Cancer Study Group: Translational bIomarker Driven UMbrella Project for Head and Neck (TRIUMPH), Esophageal Squamous Cell Carcinoma- Part 1 (HNSCC)]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Cancer Study Group (Other); Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KCSG-TRIUMPH
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: HNSCC; Head and Neck Neoplasms
Keywords: NGS; Nanostring; Biomarker Driven Umbrella Trial; BYL719,poziotinib, abemaciclib, nintedanib; Durvalumab + Tremelimumab Combination Treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Alpelisib; HM781-36B; nintedanib; abemaciclib; durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: During or after palliative 1st line platinum based chemotherapy, we will perform prescreening NGS based molecular characterization.
  Molecular tumor board to determine characterization will be held for every patients. Once each patients have relevant genetic pathway, the patients will be allocated each treatment arm.If the patients have no relevant genetic alteration, such a patients will allocated to durvalumab+/- tremelimumab arm regardeless of PD-L1 positivity. If the patients who allocated to BYL719(Arm1),poziotinib(Arm2), nintedanib(Arm3), and abemaciclib(Arm4) experience disease progression but still meet the inclusion/ exclusion criteria for durvalumab+/- tremelimumab arm((Arm5) the cross over to durvalumab+/- tremelimumab arm will be permitted. Vice versa (cross over from durvalumab+/- tremelimumab arm to another arms) is not permitted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm1: BYL719 (Experimental): Experimental: BYL719 BYL719 is an oral class I α-specific PI3K inhibitor belonging to the 2-aminothiazole class of compounds.
  Interventions: Drug: BYL719
- Arm2: Poziotinib (Experimental): Experimental:Poziotinib Poziotinib is a pan-HER tyrosine kinase inhibitor.(oral class)
  Interventions: Drug: Poziotinib
- Arm3: Nintedanib (Experimental): Nintedanib is a potent small molecule triple receptor tyrosine kinase inhibitor (PDGFR, FGFR 1-3,VEGFR 1-3 ,VEGFR- 2) is considered to be the crucial receptor involved in initiation of the formation as well as the maintenance of tumour vasculature.(oral class)
  Interventions: Drug: Nintedanib
- Arm4: Abemaciclib (Experimental): Abemaciclib represents a selective and potent small molecule CDK4 and CDK6 dual inhibitor with broad antitumor activity in preclinical pharmacology models.(oral class)
  Interventions: Drug: Abemaciclib
- Arm5: Durvalumab,Tremelimumab (Experimental): Durvalumab is a human immunoglobulin (Ig) G1 kappa (IgG1κ) monoclonal antibody (mAb) that blocks the interaction of PD-L1 with PD-1 on T-cells and CD80 on immune cells and is engineered to reduce antibody-dependent cell-mediated cytotoxicity.(IV class)
  Tremelimumab is specific for human CTLA-4; cluster of differentiation a cell surface receptor that is expressed primarily on activated T cells and acts to inhibit their activation.(IV class)
  Interventions: Drug: Durvalumab,Tremelimumab

INTERVENTIONS:
Drug: BYL719 — Patients will be instructed to take BYL719 orally at a dose of 100 mg with a glass of water once daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day.
  Arms: Arm1: BYL719
Drug: Poziotinib — Patients will be instructed to take BYL719 orally at a dose of 12 mg once daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day.
  Arms: Arm2: Poziotinib
Drug: Nintedanib — Initial dose 200 mg twice per day orally according to study protocol.
  Arms: Arm3: Nintedanib
Drug: Abemaciclib — Patients will be instructed to take Abemaciclib orally at a dose of 200mg bid with a glass of water twice daily, in a fasting state or with a light fat-free meal, and as close as possible to the same time each day.
  Arms: Arm4: Abemaciclib
Drug: Durvalumab,Tremelimumab — Durvalumab: 1.5g Q4W plusTremelimumab: 75mg Q4W up to 4cycle then Durvalumab 750mg Q2W, till PD or unacceptable toxicity.
  Arms: Arm5: Durvalumab,Tremelimumab

SUMMARY:
Open, multicenter, single arm, phase II, biomarker driven umbrella trial for head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
This study will be conducted as a part of umbrella trial by Korean Cancer Study Group. The brief scheme of this umbrella trial is as follows:

R/M HNSCC 2nd line

1. PI3K inhibitor - BYL719 (from Norvatis)
2. EGFR/HER2 inhibitor - poziotinib (from Hanmi pharmaceutical)
3. FGFR inhibitor - nintedanib (from Boehringer ingelheim)
4. Cell cycle (CDK4/6) inhibitor - abemaciclib (from Lily)
5. Others- anti PD1/PD-L1 - durvalumab+/-tremelimumab (from AZ)

During or after palliative 1st line platinum based chemotherapy, we will perform prescreening NGS based molecular characterization. The molecular characterization will be done by following three methods.

* NGS : Agilent SureSelect Target Enrichment (245 genes)
* Nanostring nCounter including immune signature
* IHC : PD-L1, CD8 TIL, p16

Mutation will be analyzed by NGS, fusion and amplification will be determined by Nanostring methods, and PD-L1/p16 status will be determined by immunohistopathology. Molecular tumor board to determine characterization will be held for every patients. Once each patients have relevant genetic pathway, the patients will be allocated each treatment arm (see below figure). If the patients have no relevant genetic alteration, such a patients will allocated to durvalumab+/- tremelimumab arm regardeless of PD-L1 positivity. If the patients who allocated to poziotinib, BYL719, nintedanib, and abemaciclib experience disease progression but still meet the inclusion/ exclusion criteria for durvalumab+/- tremelimumab arm, the cross over to durvalumab+/- tremelimumab arm will be permitted. Vice versa (cross over from durvalumab+/- tremelimumab arm to another arms) is not permitted.

ELIGIBILITY:
Common Inclusion Criteria: The following criteria must all be met.

* Histologically or cytologically confirmed recurrent or metastatic SCCHN
* Ineligibility for local therapy (surgery or radiation for curative intent)
* Prior palliative chemotherapy including platinum-based chemotherapy. When recurred within 6 months of definitive/neoadjuvant/adjuvant chemo- or chemoradiation, the chemotherapy is considered a line of palliative chemotherapyAt least one measurable lesion by RECIST ver 1.1
* Age ≥20
* ECOG performance status of 0-1
* Adequate organ function for treatment

  * Absolute neutrophil count (ANC) ≥1500 cells/mm3
  * Platelets ≥100,000 cells/mm3
  * Hemoglobin ≥ 9 g/dL.
  * Serum creatinine <1.5 x institution upper limit of normal
  * Bilirubin ≤1.5 x upper limit of normal (ULN)
  * AST (SGOT) ≤3.0 x ULN
  * ALT (SGPT) ≤3.0 x ULN
* At least one lesion that is measurable according to the RECIST 1.1 criteria by CT or MRI
* The patient has provided signed informed consent and has a compliance to follow the study protocol.

Common Inclusion Criteria: Patients eligible for this study should not meet any of the following criteria:

* Nasopharyngeal carcinoma
* Major surgery within 4 weeks prior to initiating study treatment
* Patients who have received prior systemic chemotherapy, immunotherapy or study drug within 4 weeks (Exclusion of conventional radiotherapy for non-target lesions within 2 weeks prior to enrollment)
* Pregnant woman, Breast-feeding woman
* Females who were not screened for pregnancy or had positive results. (Women are considered post-menopausal and not of child bearing potential if they have had 12 months of amenorrhea or have had surgical bilateral oophorectomy or Age ≥60
* Previous or concomitant malignant disease, except adequately treated basal cell cancer of the skin or cervical cancer in situ, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior study entry
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial (infection/inflammation, intestinal obstruction, social/psychological complications)
* Patients with significant cardiovascular disease or within AMI 12 months, (Congestive heart failure or Any significant ventricular arrhythmia)
* Patients who received organ transplants requiring immunosuppressive therapy
* Patients with HBsAg, anti-HCV, HIV-positive patients or other uncontrolled infectious diseases

  * However, Arm1-Arm3 Inactivated hepatitis B carriers using appropriate prophylactic antiviral agents can be listed at the discretion of the investigator
  * Arm5: An active HBV carrier who has received HBV DNA <100 IU / mL at the time of screening, has received appropriate prophylactic antiviral treatment and continues to receive treatment with an antiviral agent during the trial can be registered.

Specific Inclusion Exclusion Criteria: In addition to the common Inclusion / exclusion criteria, the specific drug Inclusion / exclusion criteria for the drug study should be met.

Arm 1: BYL719

BYL719 Specific Inclusion Criteria

* Patients with relevant genetic alterations including PI3K pathway alteration or those by physician's discretion based on next generation sequencing (NGS).
* Uncontrolled, untreated brain metastasis. Patients with treated/controlled and asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases ≥ 28 days (must include radiotherapy and/or surgery) and, if on corticosteroid therapy, should be receiving a stable low dose (e.g. dexamethasone 4 mg or equivalent dose of another corticosteroid for at least 14 days before start of study treatment).
* Life expectancy of at least 12 weeks

BYL719 Specific Exclusion Criteria

* Prior treatment with AKT. mTOR PI3K pathway inhibitors
* Patient who cannot take the oral drug
* Impaired GI function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration
* Clinically significant cardiac disease or impaired cardiac function, such as:

  * Congestive heart failure (CHF) requiring treatment (New Yort Heart Association (NYHA) Grade ≥ 2)
  * left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram
  * uncontrolled arterial hypertension defined by blood pressure > 140/100 mmHg at rest (average of 3 consecutive readings)
  * History or current evidence of clinically significant cardiac arrhythmias, arterial fibrillation and/or conduction abnormality, e.g. congenical long QT syndrome, high grade/complete AV-blockage
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening, QTcF> 480 msec on screening ECG
* Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with FPG ≥ 140 mg/dL/7.8mmol/L, or history of documented steroid-induced diabetes mellitus.

Arm 2: poziotinib

poziotinib Specific Inclusion Criteria

* Patients with relevant genetic alterations including EGFR/HER2 pathway alteration or those by physician's discretion based on next generation sequencing (NGS).

poziotinib Specific Exclusion Criteria

* Previous treatment with small molecule EGFR tyrosine kinase inhibitors (Cetuximab is permitted)
* Patients with uncontrolled CNS metastatic involvement. However, corticosteroids should be discontinued at least 2 weeks before clinical trials, except for radiologic and neurologically stable cases for more than 4 weeks.
* Patients with known interstitial lung disease
* Patients with uncontrolled or significant cardiovascular disease (AMI ,Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 50%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
* Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug

Arm 3: nintedanib

nintedanib Specific Inclusion Criteria

* Patients with relevant genetic alterations including FGFR athway alteration or those by physician's discretion based on next generation sequencing (NGS).
* Life expectancy of at least 12 weeks

nintedanib Specific Exclusion Criteria

* Prior treatment with FGFR pathway inhibitors
* Recent bleeding history, major vessel invasion of tumour
* Patient who cannot take the oral drug
* Patients with active brain metastases (defined as stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, or requiring treatment with anticonvulsants). Patients with treated/controlled and asymptomatic CNS metastases may participate in this trial.
* Clinically significant cardiac disease or impaired cardiac function, such as:

  * Congestive heart failure (CHF) requiring treatment (New Yort Heart Association (NYHA) Grade ≥ 2)
  * left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram
  * uncontrolled arterial hypertension defined by blood pressure > 140/100 mmHg at rest (average of 3 consecutive readings)
  * History or current evidence of clinically significant cardiac arrhythmias, arterial fibrillation and/or conduction abnormality, e.g. congenical long QT syndrome, high grade/complete AV-blockage
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening, QTcF> 480 msec on screening ECG
* Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment
* Therapeutic anticoagulation (except low-dose heparin or heparin flush in the catheter) or antiplatelet therapy (except for acetylsalicylic acid <325 mg / day)

Arm 4: abemaciclib

abemaciclib Specific Inclusion Criteria

* p16 negative and genetic alterations in CDK4/6 pathway
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to screening. A washout period of at least 21 days is required between last chemotherapy dose and screening (provided the patient did not receive radiotherapy).
* Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization

abemaciclib Specific Exclusion Criteria

* Prior treatment with CDK4/6 pathway inhibitors
* Recent significant bleeding history and major vessel invasion of tumor
* Pregnant woman, Breast-feeding woman

  * If a female of childbearing potential, must have a negative serum pregnancy test within 7 days of the first dose of abemaciclib and agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of abemaciclib.
* If a male, must agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following the last dose of abemaciclib. Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.
* The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Patient who cannot take the oral drug
* Patient who have an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies)

Arm 5: durvalumab +/- tremelimumab

durvalumab +/- tremelimumab Specific Inclusion Criteria

* NGS analysis on the molecular tumor board showed that there was no mutation corresponding to Arm 1 ~ 4 or Patients who were treated with Arm 1 ~ 4 and progressed to disease and who satisfied Arm5 criteria (Arm 1 ~ 4 allow cross over to Arm 5, but not the reverse.)

durvalumab +/- tremelimumab Specific Exclusion Criteria

* Previous treatment with CTLA-4 , PD-1 or PDL-1 inhibitors
* Symptomatic brain metastasis
* Patients with known interstitial lung disease
* Systemic immunosuppressive therapy
* Active autoimmune disease 7 - Body weight <30kg
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation
* 12-Lead electrocardiogram (ECG) with abnormal tracing or clinically significant changes that require medical intervention
* History of treatment with live vaccine within 30 days of drug administration for clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 24 months
  Arm 1: RECIST version 1.1
Response rate (RR) | 24 months
  Arm 2-5: RECIST version 1.1

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 24 months
  RECIST version 1.1
Progression-free survival (PFS) | 24 months
  RECIST version 1.1
Overall survival (OS) | 24 months
  Overall Survival is defined as the time from first dose to death due to any cause. Through the follow-up within 30 days after study completion or termination of the last subject, death and date of death will be checked for subject alive during treatment period
Time to progression (TTP) | 24 months
  RECIST version 1.1
Quality of life assessment | 24 months
  FACT-H&N (Version 4.0)
Duration of response | 24 months
  RECIST version 1.1
Toxicity: Number of patients with treatment-related AE as assessed by NCI CTCAE version 4.03 | 24 months
  number of patients with treatment-related AE as assessed by NCI CTCAE version 4.03
biomarker | 24 months
  NGS, nanostring

CONTACTS AND LOCATIONS:
Overall Officials: Hwan Jung Yun, Study Chair — Chungnam National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
anticipated as research paper

REFERENCES:
- [Derived] Keam B, Hong MH, Shin SH, Heo SG, Kim JE, Ahn HK, Lee YG, Park KU, Yun T, Lee KW, Kim SB, Lee SC, Kim MK, Cho SH, Oh SY, Park SG, Hwang S, Nam BH, Kim S, Kim HR, Yun HJ; KCSG TRIUMPH Investigators. Personalized Biomarker-Based Umbrella Trial for Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: KCSG HN 15-16 TRIUMPH Trial. J Clin Oncol. 2024 Feb 10;42(5):507-517. doi: 10.1200/JCO.22.02786. Epub 2023 Sep 12. PMID 37699162